CLINICAL TRIAL: NCT05076578
Title: A Prospective Clinical Study Evaluating the Efficiency of Full Thickness Micograft Harvesting in Healthy Volunteers and the Use of Full Thickness Micrografts in the Treatment of Patients With Chronic Wounds
Brief Title: A Prospective Clinical Study Evaluating the Harvesting of Micografts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SerenaGroup, Inc. (Network)
Collaborators: Medline Industries (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARTIST-001
Record Dates: First submitted 2021-08-27; First posted 2021-10-13 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Chronic Wound
MeSH Terms: interventions — Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: The ARTTM system is an electrically powered handheld device containing disposable sterile needle cartridges. The control elements include a push button that operates the back and forth movement of the needles in the cartridge. The device can harvest over 300 full thickness MicroColumns.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Evaluate the harvesting of micografts in healthy and patients with chronic wounds (Experimental): The ART Skin Harvesting System is intended to harvest full thickness skin microcolumns in a minimally invasive manner and scatter them at the recipient site. It consists of three components: (1) a non-sterile, reusable handheld device; (2) a sterile, single-patient use needle cartridge containing the needle array for harvesting skin micrografts from the patient donor site; and (3) a sterile, disposable handheld protective sleeve to cover the handheld device (figure 1). The sterile sleeve reduces contamination of the reusable handheld device and provides a sterile barrier between the non-sterile handheld device and the patient.
  Interventions: Device: Autologous Regeneration of Tissue (ARTTM) system

INTERVENTIONS:
Device: Autologous Regeneration of Tissue (ARTTM) system — The ART Skin Harvesting System is intended to harvest full thickness skin microcolumns in a minimally invasive manner and scatter them at the recipient site. It consists of three components: (1) a non-sterile, reusable handheld device; (2) a sterile, single-patient use needle cartridge containing the needle array for harvesting skin micrografts from the patient donor site; and (3) a sterile, disposable handheld protective sleeve to cover the handheld device (figure 1). The sterile sleeve reduces contamination of the reusable handheld device and provides a sterile barrier between the non-sterile handheld device and the patient.

SUMMARY:
ART (Autologous Regeneration of Tissue) is a revolutionary technology for harvesting skin without the drawbacks of conventional grafting. This innovative system allows the clinician to collect hundreds of microcolumns of full-thickness skin tissue and apply them directly to the wound site. It can all be done in an outpatient setting with minimized donor site concerns.

DETAILED DESCRIPTION:
Millions of Americans suffer from acute and hard-to-heal chronic wounds. The National Institutes of Health estimates that 3% of the U.S. population over the age of 65 has an open wound. As the population ages in concert with an increased incidence of diabetes and obesity, the problem will intensify. A recent article suggests that the financial burden of wound care is approaching 100 billion dollars. Despite the gravity of the problem and the number of patients afflicted, open wounds can take weeks, months or even years to heal. The search for interventions that promote healing, reduce suffering and enhance quality of life continues as does the need to address the underlying issues that disrupt the wound healing process.

Countless hours are spent treating chronic wounds (diabetic ulcers, venous ulcers, pressure injuries). Called the "silent epidemic," chronic wounds often result in infection, disability and sometimes amputation.

Crafting a treatment plan that addresses the individual needs of each wound and each patient, hinges on managing the underlying issues that can disrupt healing and increase healthcare costs. Innovation in wound bed preparation and tissue regeneration bring new hope for these patients in the form of more effective wound closure, improved quality of life and reduced costs.

Autologous skin grafting is the gold standard for covering areas of skin loss.4 However, traditional grafting is limited by accessibility issues and donor site complications-pain, risk of infection, scarring.

ART (Autologous Regeneration of Tissue) is a revolutionary technology for harvesting skin without the drawbacks of conventional grafting. This innovative system allows the clinician to collect hundreds of microcolumns of full-thickness skin tissue and apply them directly to the wound site. It can all be done in an outpatient setting with minimized donor site concerns.

ELIGIBILITY:
Inclusion Criteria:

Group A (Healthy Individuals)

1. 18 years or older.
2. Healthy participants without major diseases.

Group B (Subjects with Chronic Wounds)

1. Participants presenting with chronic wound(s) present for a minimum of 4 weeks (eg. diabetic foot ulcers (DFU), venous leg ulcers (VLU), pressure ulcers (PrU), and other acceptable etiologies).
2. 18 years or older.

Exclusion Criteria:

1. Subject on an investigational drug or therapeutic device within 30 days of the study visit.
2. Presence of a condition that PI considers will compromise the subject's ability to participate in the study.
3. Known allergy to any of the dressings or their components.
4. The subject has a history of excessive bleeding.
5. The subject has a history of keloid formation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
To evaluate wound closure | 4 weeks
  Evaluating Wound Closure with Surface area through measurments
Group A (Healthy Volunteers): The number of successful full thickness micrograft harvests from calf, thigh, and lower back as a percentage of the maximal possible grafts. | 4 weeks
  Group A (Healthy Volunteers): The number of successful full thickness micrograft harvests from calf, thigh, and lower back as a percentage of the maximal possible grafts.
Group B (Chronic Wound patients): The number of wounds achieving a percentage area reduction (PAR) of 40% or greater in 4 weeks. | 4 weeks
  Group B (Chronic Wound patients): The number of wounds achieving a percentage area reduction (PAR) of 40% or greater in 4 weeks.

SECONDARY OUTCOMES:
Proportion of patients that achieve complete wound closure | 4 weeks
  Proportion of patients that achieve complete wound closure by week 4. (Group B Only)
Time to initial wound closure within 4 weeks (Kaplan-Meier approach). | 4 weeks
  Time to initial wound closure within 4 weeks (Kaplan-Meier approach). (Group B only)
Difference in pain between baseline | 4 weeks
  Difference in pain between baseline and week 4 using a numeric scale 1-10. (Group B Only)
Number of Treatments used per patient. | 4 weeks
  Number of Treatments used per patient. (Group B Only)
• Incidence of adverse events (calculated as total and mean number per patient). | 4 weeks
  • Incidence of adverse events (calculated as total and mean number per patient). (Group B Only)

OTHER OUTCOMES:
Ease of use for the Autologous Regeneration of Tissue (ART) system using System Usability Scale (SUS). | 4 weeks
  Ease of use for the ART system using System Usability Scale (SUS).Questionnaire with a series of questions. 1 being "Strongly disagree" and 5 being "strongly agree"
Mean time required for procedure. | 4 weeks
  Mean time required for procedure.
Pain related to procedure (Group A and B). | 4 weeks
  Pain related to procedure (Group A and B) using a numeric scale 1-10.
Assess therapeutic goals and benefit using Patient Benefit Index (PBI). | 4 weeks
  Assess therapeutic goals and benefit using Patient Benefit Index (PBI).
To assess samples through blood speciman | 4 weeks
  To collect histological samples from both healthy (Group A) and non-healing patients (Group B) for hematoxylin and eosin (H&E) processing and imaging using a microscope.
To assess biopsies using the ART device. | 4 weeks
  To collect biopsies from healthy volunteerrs from H&E plus Movat and Herovici staining.
Assessing the effect of bacterial burden on wound healing using the MolecuLight Imaging Device | 4 weeks
  The effect of bacterial burden on wound healing following micrograft placement using fluorescence imaging.
Wear time of an occlusive dressing on donor site. | 4 weeks
  Wear time of an occlusive dressing on donor site.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Serena, MD,FACS, Principal Investigator — SerenaGroup, Inc.
Locations (1):
- SerenaGroup - Monroeville, Monroeville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No